CLINICAL TRIAL: NCT03448081
Title: An Exploratory, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2 Study to Evaluate the Safety, Tolerability, and Efficacy of SNA-120 (Pegcantratinib) Ointment for the Symptomatic Treatment of Persistent Pruritus and Psoriasis in Subjects Being Treated With Calcipotriene Ointment
Brief Title: Safety, Tolerability and Efficacy of SNA-120 for Treatment of Pruritus and Psoriasis in Subjects Treated With Calcipotriene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sienna Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Sienna Labs (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNA-120-202
Record Dates: First submitted 2018-02-14; First posted 2018-02-27 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pruritus; Psoriasis
MeSH Terms: conditions — Pruritus; Psoriasis | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SNA-120 + Calcipotriene (Active Comparator)
  Interventions: Drug: SNA-120; Drug: Calcipotriene
- Placebo + Calcipotriene (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Calcipotriene

INTERVENTIONS:
Drug: SNA-120 — SNA-120 (0.5%) active ointment
  Arms: SNA-120 + Calcipotriene
Drug: Placebo — Vehicle Ointment
  Arms: Placebo + Calcipotriene
Drug: Calcipotriene — Calcipotriene ointment (0.005%)

SUMMARY:
A Phase 2 study evaluating safety, tolerability, and efficacy of SNA-120 ointment when administered topically with calcipotriene ointment for the treatment of pruritus and psoriasis.

DETAILED DESCRIPTION:
All subjects are required to meet eligibility requirements and undergo a calcipotriene run-in period (Part A) prior to qualifying and randomizing into the study to receive either SNA-120 or Placebo ointment in combination with calcipotriene ointment (Part B). Combination therapy (SNA-120 ointment + calcipotriene ointment or Placebo ointment + calcipotriene ointment) is to continue over an 8 week period to evaluate safety, tolerability and the efficacy of treatment on both persistent pruritus and the visible signs and symptoms of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Stable psoriasis for at least 6 months prior to screening
* Chronic pruritus of the psoriasis plaques at least 6 weeks prior to screening
* At least moderate baseline overall itch associated with psoriatic plaques
* Willing and able to undergo a 4-week run-in with calcipotriene ointment dosing and remain on this stable regimen throughout the study
* Mild or moderate psoriasis at screening and baseline
* Subject's plaques are amenable to treatment with a topical medication
* Willing and able to discontinue all other topical products to treat psoriasis and/or itch, including topical steroids
* Willing and able to avoid prolonged exposure of the designated treatment plaques to ultraviolet (UV) radiation (natural and artificial) for the duration of the study
* Women of childbearing potential must have a negative pregnancy test and must agree to use highly effective methods of contraception during the study
* Men who engage in sexual activity that can result in fathering children must agree to use highly effective forms of contraception during the study

Exclusion Criteria:

* Underlying conditions other than psoriasis that, in the opinion of the investigator, currently cause or influence pruritus of the overall skin
* Current or past history of hypercalcemia, Vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders
* Thyroid abnormalities that, in the opinion of the investigator, are clinically relevant and may affect assessments
* Current diagnosis of guttate, erythrodermic, exfoliative, or pustular psoriasis
* Subjects with a clinical diagnosis of bacterial infection of the skin
* Subjects who have previously failed treatment with or failed to tolerate treatment with calcipotriene
* Known hypersensitivity to SNA-120 (pegcantratinib), calcipotriene, the study treatment excipients, and /or polyethylene glycol (PEG), or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation
* Currently enrolled in an investigational drug or device study or has used an investigational drug or an investigational device treatment within 30 days or 5 half-lives of investigational drug (whichever is longer) of baseline
* Women who are pregnant or lactating, or are planning to become pregnant during the study
* Subjects previously participating in any SNA-120 (and/or CT327 or pegcantratinib) clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Change in Itch Numeric Rating Scale scores (I-NRS) from baseline | week 8
  11-point NRS scale used to assess pruritus severity, ranging from 0 (no itching at all) to 10 (worst possible itching)

SECONDARY OUTCOMES:
Change in Investigator Global Assessment (IGA) from baseline | week 8
  5-point scale used to assess the overall severity of psoriasis by evaluting induration, erythema and desquamation (0=clear to 4=severe)
Change in Psoriasis Area Severity Index (PASI) from baseline | week 8
  A quantitative rating score for measuring the severity of psoriatic lesions based on area coverage and plaque appearance (0 = no disease to 72 = maximum disease)

OTHER OUTCOMES:
Safety measured by frequency of Adverse Events | week 10
  Frequency of all Adverse Events (AEs), including local site reactions that occur during the trial from baseline through week 10
Safety measured by severity of Adverse Events | week 10
  Severity of all Adverse Events (AEs), including local site reactions that occur during the trial from baseline through week 10
Safety measured by change in clinical lab results from baseline | week 10
  biochemistry lab assessments
Safety measured by change in clinical lab results from baseline | week 10
  Clinical laboratory assessments include urinalysis (pH, glucose, protein)
Safety measured by change in clinical lab results from baseline | week 10
  hematology lab assessments
Safety measured by change from baseline in blood pressure | week 10
  Systolic/diastolic blood pressure (BP in mmHg) - measured every full clinic visit, from baseline through week 10
Safety measured by change from baseline in pulse | week 10
  Measured in beats per minute (bpm) - measured every full clinic visit, from baseline through week 10
Safety measured by number of abnormal physical examinations from baseline | week 8
Safety measured by PR/PQ intervals measured by 12-lead ECG | week -4
  Safety measured by PR/PQ intervals measured by 12-lead ECG at screening
Safety measured by PR/PQ intervals measured by 12-lead ECG | week 0
  Safety measured by PR/PQ intervals measured by 12-lead ECG at baseline
Safety measured by PR/PQ intervals measured by 12-lead ECG | week 4
  Safety measured by PR/PQ intervals measured by 12-lead ECG at week 4
Safety measured by PR/PQ intervals measured by 12-lead ECG | week 8
  Safety measured by PR/PQ intervals measured by 12-lead ECG at week 8
Safety measured by QRS duration measured by 12-lead ECG | week -4
  Safety measured by QRS duration measured by 12-lead ECG at screening
Safety measured by QRS duration measured by 12-lead ECG | week 0
  Safety measured by QRS duration measured by 12-lead ECG at baseline
Safety measured by QRS duration measured by 12-lead ECG | week 4
  Safety measured by QRS duration measured by 12-lead ECG at week 4
Safety measured by QRS duration measured by 12-lead ECG | week 8
  Safety measured by QRS duration measured by 12-lead ECG at week 8
Safety measured by QT intervals measured by 12-lead ECG | week -4
  Safety measured by QT intervals measured by 12-lead ECG at screening
Safety measured by QT intervals measured by 12-lead ECG | week 0
  Safety measured by QT intervals measured by 12-lead ECG at baseline
Safety measured by QT intervals measured by 12-lead ECG | week 4
  Safety measured by QT intervals measured by 12-lead ECG at week 4
Safety measured by QT intervals measured by 12-lead ECG | week 8
  Safety measured by QT intervals measured by 12-lead ECG at week 8

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Sienna 018, Anniston, Alabama
  - Sienna 009, Mobile, Alabama
  - Sienna 019, Fountain Valley, California
  - Sienna 007, Los Angeles, California
  - Site 016, Sherman Oaks, California
  - Site 013, Coral Gables, Florida
  - Site 015, Sanford, Florida
  - Site 012, Indianapolis, Indiana
  - Sienna 011, Warren, Michigan
  - Sienna 005, Berlin, New Jersey
  - Sienna 020, Rochester, New York
  - Site 014, Raleigh, North Carolina
  - Sienna 002, Oklahoma City, Oklahoma
  - Sienna 017, Austin, Texas
  - Sienna 010, Houston, Texas
  - Sienna 021, Pflugerville, Texas
  - Sienna 001, San Antonio, Texas
- Canada (3):
  - Sienna 006, Surrey, British Columbia
  - Sienna 008, Peterborough, Ontario
  - Sienna 003, Montreal, Quebec